CLINICAL TRIAL: NCT05845697
Title: Immediate Effect of Dry Needling of the Lumbar Multifidus on Pain Sensitivity In A Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202202632
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain
Keywords: trigger point dry needling; quantitative sensory testing; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Double blind, randomized control
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actual dry needling group (Experimental): Will receive actual dry needling of the lumbar multifidus with a 50-60mm filiform needle
  Interventions: Other: Trigger point dry needling
- Sham dry needling group (Sham Comparator): Will receive needling from a sham needle that is blunted so it does not pierce the skin but has been shown to be valid for being indistinguishable from receiving an actual needle.
  Interventions: Other: Sham dry needling

INTERVENTIONS:
Other: Trigger point dry needling — Filiform needle that pierces the skin and is inserted into an identified trigger point in the muscle
  Arms: Actual dry needling group
Other: Sham dry needling — A validated sham dry needle that is blunted on the end and does not pierce the skin
  Arms: Sham dry needling group

SUMMARY:
The goal of this interventional study is to test the effects of trigger point dry needling to the low back in a healthy population. The main aims are to answer:

* Is there a change in sensitivity to experimental pain after trigger point dry needling
* To determine if there is an association between demographic and psychological factors and immediate changes in pain sensitivity after receiving trigger point dry needling.

Participants will be randomly assigned to one of two groups a dry needling group or a sham dry needling group. The dry needling group will receive trigger point dry needling to the lumbar spine. The sham dry needling group will receive needling to the lumbar spine with a sham needle which does not penetrate the skin.

In other words, researchers will compare an intervention group and a sham group to see if dry needling has an immediate change in pain sensitivity in response to experimentally induced pain.

DETAILED DESCRIPTION:
The intent of this study is to investigate the effects of trigger point dry needling on pain sensitivity in a healthy population. In this study, the effects of trigger point dry needling will be measured using quantitative sensory testing. This is a method of testing pain sensitivity by providing a painful stimulus and having the participant rate their response to the stimulus on a pain scale. In this way, the researchers will be able to determine changes to participant's response to painful stimuli and changes to the nervous system after trigger point dry needling interventions to the low back. This information will provide important insight as to how dry needling modulates pain.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 65
* Be pain-free

Exclusion Criteria:

* Participants will not be excluded on the basis of race or gender but will be excluded if they meet any of the following exclusion criteria:
* a) Non-English speaker
* b) presence of a medical condition known to affect sensation
* c) history of surgery to the low back
* d) history of blood clotting disorders or medical conditions associated with bleeding disorders
* e) Current use of the medication causing difficulty with clotting (such as blood thinners)
* f) Contraindication to the application of needles including, but not limited to, fear of needles or metal allergy --g) women who are pregnant or planning on becoming pregnant any contraindication to application of ice or cold pack, such as: uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, and circulatory compromise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-13 (Actual)

PRIMARY OUTCOMES:
Change in Heat Thermal Pain Threshold degrees Celsius baseline and Heat Thermal Pain Threshold degrees Celsius immediately following intervention | Baseline and immediately following the intervention
  Participants will indicate when an thermode of ascending temperatures first changes from a sensation of warmth to painful by saying "pain" and indicating the amount of pain with a visual analog scale. This change will be calculated by taking the difference between the two scores.
Change in Cold Thermal Pain Threshold degrees Celsius baseline and Cold Thermal Pain Threshold degrees Celsius immediately following intervention | Baseline and immediately following the intervention
  Participants will indicate when an thermode of descending temperatures first changes from a sensation of cold to painful by saying "pain" and indicating the amount of pain with a visual analog scale. This change will be calculated by taking the difference between the two scores.
Change in Pressure Pain Threshold Kilopascals baseline and Pressure Pain Threshold Kilopascals immediately after following intervention | Baseline and immediately following the intervention
  Participants will indicate when ascending pressure from an algometer first changes from a sensation of pressure to painful by saying "pain" and indicating the amount of pain with a visual analog scale. This change will be calculated by taking the difference between the two scores.
Change in baseline Thermal Temporal Summation | Baseline and immediately following the intervention
  Participants will rate the pain associated with a series of 10 heat pulses applied to the skin on a 0 to 100 numerical rating scale with 0= no pain to 100= worst pain imaginable.
Change in baseline After sensation | Baseline and immediately following the intervention
  After sensation is the term used to describe the measurement of pain that remains after a painful stimulus.
  Participants will rate the pain remaining every 15 seconds for a total of one minute following the final thermal pulse in the Thermal Temporal Summation protocol (as described in outcomes 4). The numeric rating scale is (0 - 100) with "0" being no pain at all and "100" being worst pain imaginable
Change in baseline Conditioned pain modulation | Baseline and immediately following the intervention
  Pressure pain threshold will be assessed immediately prior to and following a pain inducing cold water bath immersion. Condition pain modulation will be defined by the changes in pressure pain threshold prior to and immediately following the cold water bath immersion

SECONDARY OUTCOMES:
Expectations | Baseline, immediately following intervention
  Expectation will be assessed using a 15 point global rating of change anchored with -7= expect a very great deal more pain; 0= unchanged, and 7= a very great deal less pain
Degree to which expectations met | Immediately following follow pain testing
  Single question, In response to the pain testing, participants will be asked to indicate, "How would you describe how you feel now compared to how you expected" categorically, with "more", "less", or "expected" level of pain
Blinding | Immediately following the assigned intervention
  Five point scale with 1= "strongly believe the treatment is active" and 3= "somewhat believe the treatment is placebo" and 5= "do not know"

CONTACTS AND LOCATIONS:
Overall Officials: Joel Bialosky, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No